CLINICAL TRIAL: NCT03430817
Title: Citicholine-Amantadine Trial in Traumatic Brain Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dina Salah Eldin Mahmoud Badre, Assistant Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU R44/2017
Record Dates: First submitted 2018-01-05; First posted 2018-02-13 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Intensive Care Unit
MeSH Terms: interventions — Cytidine Diphosphate Choline; Amantadine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group C (Experimental): Citicholine Drug
  Interventions: Drug: Citicholine
- Group A (Experimental): Amantadine Drug
  Interventions: Drug: Amantadine
- Group D (Experimental): Both Citocholine and Amantadine
  Interventions: Drug: Citicholine; Drug: Amantadine

INTERVENTIONS:
Drug: Citicholine — Patients will receive 1 gram (2 vials of citicholine; each 500 mg) every 12 hours given slowly intravenous over 10 minutes for 7 days then oral form of the drug will be used. Participants who can swallow will receive 500-mg (5ml volume; 100mg/ml) oral drops (syrup) twice a day. Participants who cannot swallow will receive the same dose as oral drops syrup of citicoline through a nasogastric (NG) tube or percutaneous endoscopic gastrostomy (PEG) tube in a total dose of 1000 mg/day for the remainder of the 30 days study period.
  Arms: Group C; Group D
Drug: Amantadine — Patients will receive 200 mg of amantadine sulphate in a 500 ml solution every 12 hours by slow intravenous infusion over a period of 4 hours for 7 days then oral form will be used. Participants who can swallow will receive two 100-mg tablets twice a day. Participants who cannot swallow will receive the tablets of amantadine through a NG tube or PEG tube as 400 mg via crushed tablets with a 25-mL saline or water flush for the remainder of the 30 days study period.
  Arms: Group A; Group D

SUMMARY:
This randomized study aims at comparing between the effects of amantadine, citcholine and its combinations on arousal and behavioral consequences in early phase of moderate Traumatic Brain injury (TBI).

DETAILED DESCRIPTION:
As both agents amantadine and citcholine showed considerable effects on neuro-recovery from TBI, The investigators hypothesized that combination therapy of both drugs will have significant effect as it simultaneously will target multiple mechanisms of injury. So, this randomized study aims at comparing between the effects of amantadine, citcholine and their combinations on arousal and behavioral consequences in early phase of moderate TBI

ELIGIBILITY:
Inclusion Criteria:

* Sustained moderate non-penetrating TBI with GCS of 9-12

Exclusion Criteria:

* Patients with mild (GCS > 12) or severe TBI (GCS < 9)
* Patients suffering from any central nervous system disability prior to the traumatic brain injury
* Major medical problems as; major cardiovascular disease or heart failure, renal insufficiency (creatinine clearance, less than 60 ml per minute), liver impairment,
* Pregnancy,
* More than one seizure in the previous month,
* Prior treatment with amantadine,
* Allergy to the study drugs.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2024-03-24 (Actual); Study Completion 2024-04-20 (Actual)

PRIMARY OUTCOMES:
Galsgow coma scale | 30 days
  Neurological scale which aims to give a reliable and objective way of recording the conscious state of a person for initial as well as subsequent assessment. A patient is assessed against the criteria of the scale, and the resulting points give a patient score between 3 (indicating deep unconsciousness) and 15 (full conscious).

SECONDARY OUTCOMES:
disability rating scale (DRS) | 30 days
  The Disability Rating Scale (DRS) was developed and tested with older juvenile and adult individuals with moderate and severe traumatic brain injury (TBI). The maximum score a patient can obtain on the DRS is 29 (extreme vegetative state). A person without disability would score zero. The DRS rating must be reliable, i.e., obtained while the individual is not under the influence of anesthesia, other mind-altering drugs, recent seizure, or recovering from surgical anesthesia.
Mini Mental scale (MMS) | 30 days
  The Mini-Mental State Examination (MMSE) is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment.
  Any score greater than or equal to 24 points (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No